CLINICAL TRIAL: NCT03296241
Title: Non-ablative Er:Yttrium Aluminum Garnet (Er:YAG) Laser Therapy Effect on Stress Urinary Incontinence (SUI) Related Quality of Life and Sexual Function: a Randomized Controlled Trial
Brief Title: Non-ablative Er:Yttrium Aluminum Garnet Laser for Stress Urinary Incontinence (SUI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Adolf Lukanovič (Other)
Responsible Party: Sponsor-Investigator, Dr Adolf Lukanovič, Medical Director of the Division of Gynecology, University Medical Centre Ljubljana
Organization: University Medical Centre Ljubljana (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SUI_ErYAG_Sham
Record Dates: First submitted 2017-09-21; First posted 2017-09-28 (Actual); Last update posted 2017-09-28 (Actual); Status verified 2017-09

CONDITIONS: Stress Urinary Incontinence
Keywords: stress urinary incontinence; sexual dysfunction; laser; Er:YAG; vaginal laser; vaginal tightening; non-ablative; minimally-invasive
MeSH Terms: conditions — Urinary Incontinence, Stress; Sexual Dysfunction, Physiological | interventions — Lasers

STUDY DESIGN:
Intervention Model Description: Patients assigned randomly to two groups: laser-treatment group and sham (control) group
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients are unaware of the assignment. Both groups were treated according to the IncontiLaseTM clinical treatment protocol for SUI with non-ablative thermal-only Er:YAG laser, except that there was no energy output when treating the sham group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser (Experimental): One session of non-ablative Er:YAG laser (2940 nm) treatment of the vaginal wall, introitus and vestibule.
  Interventions: Device: laser
- Sham control (Sham Comparator): The sham control group was treated with the same procedure but with zero intensity settings - without receiving therapeutic irradiation (placebo).
  Interventions: Device: sham control

INTERVENTIONS:
Device: laser
  Other Names: IncontiLaseTM; IncontiLase
  Arms: Laser
Device: sham control
  Other Names: placebo
  Arms: Sham control

SUMMARY:
Stress urinary incontinence (SUI) is a common complaint in women after childbirth. The aim of this study was to evaluate the efficacy and safety of non-ablative Er:YAG laser therapy in the treatment of SUI and improvement of sexual gratification in parous women. 114 premenopausal parous women with SUI were randomized in two groups of 57 women; a laser intervention group and sham control (placebo) group. Both groups were treated according to the IncontiLaseTM clinical treatment protocol for SUI with non-ablative thermal-only Er:YAG laser, except that there was no energy output when treating the sham group. Patients were blinded to the allocation. At baseline and 3 months after treatment patients were clinically examined, answered questionnaires for SUI severity sexual function assessment and their pelvic floor muscle (PFM) function was assessed with perineometry. The improvement in the laser group will be compared to the improvement in the sham group.

DETAILED DESCRIPTION:
Stress urinary incontinence (SUI) is a common complaint in women after childbirth. It affects their quality of life and sexual satisfaction and is one of the major reasons for gynaecological surgery. There is a need for effective non-invasive treatment alternatives. The aim of this study was to evaluate the efficacy and safety of non-ablative Er:YAG laser therapy in the treatment of SUI and improvement of sexual gratification in parous women. 114 premenopausal parous women with SUI were randomized in two groups of 57 women; a laser intervention group and sham control (placebo) group. Both groups were treated according to the IncontiLaseTM clinical treatment protocol for SUI with non-ablative thermal-only Er:YAG laser, except that there was no energy output when treating the sham group. Patients were blinded to the allocation. At baseline and 3 months after treatment patients were clinically examined, answered questionnaires for SUI severity sexual function assessment and their pelvic floor muscle (PFM) function was assessed with perineometry. Validated International Consultation on Incontinence Questionnaire - Urinary Incontinence Short Form (ICIQ-UI SF) was used as the primary outcome measure. The Pelvic Organ Prolapse Urinary Incontinence Sexual Questionnaire short form (PISQ-12) and The Female Sexual Function Index (FSFI) were used to assess the sexual function. Patients were monitored for discomfort and side-effects during treatment and follow up period.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of stress urinary incontinence
* sexually active
* at least one vaginal delivery

Exclusion Criteria:

* pelvic organ prolapse greater than stage I
* urgency or mixed UI
* infection
* previous gynaecologic surgery or irradiation
* refuse consent

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2012-08-01 (Actual); Primary Completion 2013-08-30 (Actual); Study Completion 2013-08-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in ICIQ-UI SF score | at 3 months after intervention
  International Consultation on Incontinence Questionnaire - Urinary Incontinence Short Form

SECONDARY OUTCOMES:
Change from baseline in PISQ-12 score | at 3 months after intervention
  The Pelvic Organ Prolapse Urinary Incontinence Sexual Questionnaire
Change from baseline in FSFI score | at 3 months after intervention
  The Female Sexual Function Index, a validated generalized questionnaire utilized to assess sexual function in women in a general population.
Change from baseline in perineometry variable maximal contraction pressure | at 3 months after intervention
  Measured with Myomed 632 perineometer with the women in supine position.
Change from baseline in perineometry variable average contraction pressure | at 3 months after intervention
  Measured with Myomed 632 perineometer with the women in supine position.
Change from baseline in perineometry variable mean muscle endurance (stamina) | at 3 months after intervention
  Measured with Myomed 632 perineometer with the women in supine position.

OTHER OUTCOMES:
Side effects | up to 3 months after intervention
  Monitoring for side effects during and after intervention

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ippolito GM, Crescenze IM, Sitto H, Palanjian RR, Raza D, Barboglio Romo P, Wallace SA, Orozco Leal G, Clemens JQ, Dahm P, Gupta P. Vaginal lasers for treating stress urinary incontinence in women. Cochrane Database Syst Rev. 2025 Jul 25;7(7):CD013643. doi: 10.1002/14651858.CD013643.pub2. PMID 40709601